CLINICAL TRIAL: NCT04062045
Title: Efficacy of Continous Regional Anesthesia Using m. Erector Spinae Catheter After Video-assisted Thoracic Surgery Procedures
Brief Title: Efficacy of Continous Regional Anesthesia Using m. Erector Spinae Catheter After VATS Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Surgery Bitenc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0120- 372/2019
Record Dates: First submitted 2019-08-18; First posted 2019-08-20 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Neoplasm of Lung; Thoracic Surgery, Video-Assisted
Keywords: Anesthesia, Conduction
MeSH Terms: conditions — Lung Neoplasms | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: Masking the infusion mixture by using the same shape of the drug/placebo bottle and wrapping it into non-transparent sheath.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Local anesthetic group (Experimental): Group A will receive a continuous infusion of ropivacaine 0,2% 5ml/h and intermittent boluses of the same local anesthetic 15ml/4h through the erector spinae catheter.
  Interventions: Drug: Ropivacaine Hcl 0.2% Inj Vil 10Ml
- Group B - Placebo group (Placebo Comparator): Group B will receive a continuous infusion of 0,9% saline 5ml/h and intermittent boluses of the same fluid 15ml/4h through the erector spinae catheter.
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Ropivacaine Hcl 0.2% Inj Vil 10Ml — Group A will receive the medicine through the erector spinae catheter.
  Arms: Group A - Local anesthetic group
Drug: Saline 0.9% — Group B will receive Saline 0,9% through the erector spinae catheter.
  Arms: Group B - Placebo group

SUMMARY:
Investigators will analyze the efficacy of continuous regional anesthesia through a catheter under erector spinae muscle in a prospective, randomized, double blind, placebo-controlled study. Investigators will include 50 adults, predicted for elective lung surgery with video-assisted thoracic surgery (VATS) technique. Patients will be randomly assigned to group A or B.

Investigators will insert a catheter under the erector spinae muscle (ESC) at the T4 level of the operated side under ultrasound guidance. All patients will receive an initial bolus of 20ml levobupivacaine 0,5% through the catheter. Group A will receive a continuous infusion 5ml/h of ropivacaine 0,2% and intermittent boluses of the same local anesthetic 15ml/4h through the ESC. Group B will receive a continuous infusion of 0,9% saline in the same doses. All patients will have a PCA pump with piritramide 1mg/ml to cover the pain. All patients will receive regular doses of paracetamol and metamizole as part of multimodal analgesia.

Investigators will compare pain, assessed with the VAS scale in resting and coughing and piritramide usage in both groups. Investigators will compare the incentive spirometry results at 24 and 48 hours postoperatively and observe for possible late complications.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* ASA I-III
* Elective video-assisted thoracic surgery with 3 ports technique
* No contraindications for regional anesthesia

Exclusion Criteria:

* Allergy to local anesthetic
* Pregnancy, breastfeeding
* BMI>35
* Inflammation in the area of ES catheter insertion
* Inability to use the PCA pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Usage of opioid analgetics | Continually 48 hours post surgery
  Investigators will measure the total consumption of i.v. piritramide after surgery.

SECONDARY OUTCOMES:
Subjective pain score | Every hour in the 48 hours post surgery
  Investigators will measure subjective perception of pain with the visual analogue scale (VAS) scoring system at resting and coughing. The VAS scoring system is a numerical scale from 0-10, with 0 being no pain and 10 the strongest pain imaginable. Patients will assess their pain with the help of analogue scale with colours and faces by each number representing different VAS pain levels.
Incentive spirometry | 24 and 48 hours after surgery
  Investigators will assess spirometry with a manual device.
Satisfaction with analgesia | 1 day (at dismissal from hospital.)
  Investigators will assess satisfaction with qualitative and quantitative questionnaries.

OTHER OUTCOMES:
Complications | 2 months
  Investigators will follow up the patients in weeks after surgery for possible complications.

CONTACTS AND LOCATIONS:
Overall Officials: Polona Gams, MD, Principal Investigator — Surgery Bitenc
Locations (1):
- Surgery Bitenc, Golnik, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Anonymous IPD may be shared.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After the collection of data has finished.
Access Criteria: Primary researcher consent.

REFERENCES:
- [Background] Ahmed Z, Samad K, Ullah H. Role of intercostal nerve block in reducing postoperative pain following video-assisted thoracoscopy: A randomized controlled trial. Saudi J Anaesth. 2017 Jan-Mar;11(1):54-57. doi: 10.4103/1658-354X.197342. PMID 28217054
- [Background] Bialka S, Copik M, Daszkiewicz A, Rivas E, Ruetzler K, Szarpak L, Misiolek H. Comparison of different methods of postoperative analgesia after thoracotomy-a randomized controlled trial. J Thorac Dis. 2018 Aug;10(8):4874-4882. doi: 10.21037/jtd.2018.07.88. PMID 30233861
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] de Haan JB, Hernandez N, Sen S. Erector spinae block for postoperative analgesia following axillary hidradenitis suppurativa resection: a case report. Local Reg Anesth. 2018 Nov 15;11:87-90. doi: 10.2147/LRA.S179830. eCollection 2018. PMID 30532584
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005
- [Background] Singh S, Choudhary NK, Lalin D, Verma VK. Bilateral Ultrasound-guided Erector Spinae Plane Block for Postoperative Analgesia in Lumbar Spine Surgery: A Randomized Control Trial. J Neurosurg Anesthesiol. 2020 Oct;32(4):330-334. doi: 10.1097/ANA.0000000000000603. PMID 31033625
- [Background] Yayik AM, Cesur S, Ozturk F, Ahiskalioglu A, Ay AN, Celik EC, Karaavci NC. Postoperative Analgesic Efficacy of the Ultrasound-Guided Erector Spinae Plane Block in Patients Undergoing Lumbar Spinal Decompression Surgery: A Randomized Controlled Study. World Neurosurg. 2019 Jun;126:e779-e785. doi: 10.1016/j.wneu.2019.02.149. Epub 2019 Mar 8. PMID 30853517
- [Background] Tulgar S, Senturk O. Ultrasound guided Erector Spinae Plane block at L-4 transverse process level provides effective postoperative analgesia for total hip arthroplasty. J Clin Anesth. 2018 Feb;44:68. doi: 10.1016/j.jclinane.2017.11.006. Epub 2017 Nov 14. No abstract available. PMID 29149734
- [Background] Scimia P, Basso Ricci E, Droghetti A, Fusco P. The Ultrasound-Guided Continuous Erector Spinae Plane Block for Postoperative Analgesia in Video-Assisted Thoracoscopic Lobectomy. Reg Anesth Pain Med. 2017 Jul/Aug;42(4):537. doi: 10.1097/AAP.0000000000000616. No abstract available. PMID 28632673
- [Background] Yenidunya O, Bircan HY, Altun D, Caymaz I, Demirag A, Turkoz A. Anesthesia management with ultrasound-guided thoracic paravertebral block for donor nephrectomy: A prospective randomized study. J Clin Anesth. 2017 Feb;37:1-6. doi: 10.1016/j.jclinane.2016.10.038. Epub 2016 Dec 15. PMID 28235492
- [Background] Helms O, Mariano J, Hentz JG, Santelmo N, Falcoz PE, Massard G, Steib A. Intra-operative paravertebral block for postoperative analgesia in thoracotomy patients: a randomized, double-blind, placebo-controlled study. Eur J Cardiothorac Surg. 2011 Oct;40(4):902-6. doi: 10.1016/j.ejcts.2011.01.067. Epub 2011 Mar 5. PMID 21377888
- [Background] Hong B, Bang S, Chung W, Yoo S, Chung J, Kim S. Multimodal analgesia with multiple intermittent doses of erector spinae plane block through a catheter after total mastectomy: a retrospective observational study. Korean J Pain. 2019 Jul 1;32(3):206-214. doi: 10.3344/kjp.2019.32.3.206. PMID 31257829
- [Background] Kwon WJ, Bang SU, Sun WY. Erector Spinae Plane Block for Effective Analgesia after Total Mastectomy with Sentinel or Axillary Lymph Node Dissection: a Report of Three Cases. J Korean Med Sci. 2018 Nov 5;33(45):e291. doi: 10.3346/jkms.2018.33.e291. No abstract available. PMID 31044575
- [Background] Kot P, Rodriguez P, Granell M, Cano B, Rovira L, Morales J, Broseta A, Andres J. The erector spinae plane block: a narrative review. Korean J Anesthesiol. 2019 Jun;72(3):209-220. doi: 10.4097/kja.d.19.00012. Epub 2019 Mar 19. PMID 30886130
- [Background] Piccioni F, Ragazzi R. Anesthesia and analgesia: how does the role of anesthetists changes in the ERAS program for VATS lobectomy. J Vis Surg. 2018 Jan 11;4:9. doi: 10.21037/jovs.2017.12.11. eCollection 2018. PMID 29445595
- [Background] Luis-Navarro JC, Seda-Guzman M, Luis-Moreno C, Lopez-Romero JL. The erector spinae plane block in 4 cases of video-assisted thoracic surgery. Rev Esp Anestesiol Reanim (Engl Ed). 2018 Apr;65(4):204-208. doi: 10.1016/j.redar.2017.12.004. Epub 2018 Jan 11. English, Spanish. PMID 29336785
- [Background] Ince I, Ozmen O, Aksoy M, Zeren S, Ulas AB, Aydin Y. Erector Spinae Plane Block Catheter Insertion under Ultrasound Guidance for Thoracic Surgery: Case Series of Three Patients. Eurasian J Med. 2018 Oct;50(3):204-206. doi: 10.5152/eurasianjmed.2018.18147. PMID 30515044